CLINICAL TRIAL: NCT04139330
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Parallel Group Trial to Investigate the Proof of Concept of NPC-06 to Acute Pain in Herpes Zoster
Brief Title: NPC-06 to Acute Pain in Herpes Zoster
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NPC-06-5
Record Dates: First submitted 2019-10-18; First posted 2019-10-25 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2020-06

CONDITIONS: Acute Pain in Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NPC-06 (high dose) (Experimental): Infuse diluted NPC-06 18mg/kg solution with 3 to 4 times volume of saline. Administarate NPC-06 gradually (slowly) over 18 minutes.
  Interventions: Drug: NPC-06
- NPC-06 (low dose) (Experimental): Infuse diluted NPC-06 12mg/kg solution with 3 to 4 times volume of saline. Administarate NPC-06 gradually (slowly) over 12 minutes
  Interventions: Drug: NPC-06
- NPC-06 (placebo) (Placebo Comparator): Infuse NPC-06 (placebo) over 12 minutes or 18 minutes
  Interventions: Drug: NPC-06

INTERVENTIONS:
Drug: NPC-06 — Infuse NPC-06 intravenously

SUMMARY:
The purpose of this trial is to investigate the efficiency of pain relief and the safety of NPC-06 for the acute pain in herpes zoster in the placebo-controlled double-blind parallel group trial, in addition to explore the effective concentration of NPC-06.

DETAILED DESCRIPTION:
The eligible patients will be randomized into three groups, and will receive single doses of NPC-06 (high dose and low dose) or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. 20 years old or over at the time of informed consent.
2. Both genders.
3. Patients who have acute rash (either erythema or papule or bulla or pustule, or more), except who have crust more than 20% of entire rash at just before the time of the first administration.
4. Patients who are administrated antiviral drug for herpes zoster at the time of the first administration.
5. Patients who are administrated non-opioid analgesics(acetaminophen, NSAIDs) for herpes zoster at the time of the first administration.
6. Patients who the NRS score at the time of below evaluation point is higher than 4.

   * 120 minutes before the start of infusion.
   * Just before the start of infusion.
7. Patients who the therapeutic effect of non-opioid analgesics for herpes zoster has been insufficient.
8. Patients who can admit to hospital for the all assessment duration from first administration until next day (including hospitalized patient).
9. Patients or his/her guardian who give a written informed consent in understanding and willingness after having received enough explanation regarding the study participation.

Exclusion Criteria:

1. Patients who cannot evaluate NRS by themselves.
2. Patients who are suspected to intracranial pressure increase.
3. Patients who have epilepsy, serious psychiatric or serious neurological disease (i. e. dementia, Parkinson disease and schizophrenic disorder) or consciousness disorder.
4. Patients who have malignant tumors (except for patients who have no signs of recurrence under treatment) or patients who are under treatment for HIV or patients who are receiving immunosuppressant.
5. Patients who have complicated idiopathic trigeminal neuralgia.
6. Patients who have other serious pain which may affect the evaluation of acute herpetic pain.
7. Patients who are receiving opioids or steroids(systemic).
8. Patients who have sinus bradycardia or serious disturbance of conduction system.
9. Patients who have history of hypersensitivity against hydantoin compound.
10. Patients who are receiving tadalafil (for pulmonary hypertension), rilpivirine, asunaprevir, daclatasvir, vaniprevir, macitentan or sofosbuvir.
11. Patients who are receiving medications for neuropathic pain, antidepressants, antiarrhythmic drugs, N-methyl-D-aspartate receptor antagonists, muscle relaxants, local anesthetics, an extract from inflammatory rabbit skin inoculated by vaccinia virus, Chinese herbal medications for analgesia, vitamin B12.
12. Patients who are receiving amenamevir.
13. Patients who have meningitis or meningeal irritation signs.
14. Patients who have complications such as serious heart disease, hepatic function disorder or renal function disorder which severity are considered by investigator as grade 3 or more severe with reference to ''Concerning classification criteria for seriousness of adverse drug reactions of medical agents'' .
15. Patients who are receiving fosphenytoin, phenytoin or ethotoin and combination drug including these or have taken these drugs as adjuvant therapy for pain .

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
The improvement of NRS (Numeric Rating Scale:Max10, Min0, higher scores mean a worse outcome) score | 120 minutes after first administration
  The average change (slope) of NRS score at the time of evaluation, which is measured before the first administration, 30, 60, 90 and 120 minutes after the first administration.

SECONDARY OUTCOMES:
The improvement of NRS (Numeric Rating Scale:Max10, Min0, higher scores mean a worse outcome) score | 120 minutes after first administration
  The change of NRS score at the time of evaluation compared to baseline.
The improvement of NRS (Numeric Rating Scale:Max10, Min0, higher scores mean a worse outcome) score | 120 minutes after first administration
  The ratio of subjects who improve 2 or more points compared to baseline at 120 minutes after first administration.
The improvement of QOL(EQ-5D-5L, Max 1.000, Min -0.111, higher scores mean a better outcome) score | 7 days
  The change of QOL score at the time of evaluation compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Kawasaki Hospital, Okayama, Okayama-ken, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Iseki M, Yamamoto T, Ogawa Y, Majima Y, Abe Y, Watanabe D, Amaya F, Hasegawa T, Inafuku K, Kosugi T, Nomura Y, Deguchi T, Hamada T, Shimizu K, Arai S, Takahashi M, Hamada I, Ishikawa Y, Kawashima M. Efficacy and safety of intravenous fosphenytoin for patients with acute herpes zoster-associated pain: A placebo-controlled randomized trial. J Dermatol. 2024 Feb;51(2):234-242. doi: 10.1111/1346-8138.17054. Epub 2023 Dec 27. PMID 38149403